CLINICAL TRIAL: NCT00785031
Title: Internet-based Vascular Risk Factor Management for Patients With Clinical Manifest Vascular Disease; a Randomized Controlled Trial
Brief Title: Internet Based Vascular Risk Factor Intervention and Self Management Study
Acronym: IRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, dr.Frank L.J. Visseren, Prof., UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80-00702-98-084 ZonMw; 08-119/O (Other: METC UMC Utrecht)
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Cardiovascular Diseases
Keywords: risk management; Self Management; Self-Efficacy; Disease management; nurse practitioner; internet; risk factors; vascular diseases; economic evaluation
MeSH Terms: conditions — Cardiovascular Diseases; Vascular Diseases | interventions — Disease Management; Self-Management; Nurse Practitioners; Patient Portals; Risk Factors; Primary Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- internet based intervention (Active Comparator)
  Interventions: Other: internet based vascular risk factor intervention
- usual care (No Intervention): Patients receive their usual care from their specialist or general practitioner.

INTERVENTIONS:
Other: internet based vascular risk factor intervention — The patient and a nurse practitioner create an internet dossier and the patient is instructed on how to use the internet dossier. The internet dossier is mainly meant for the patient: to improve knowledge of vascular risk factors, to give an overview of the actual status of the levels of his/her vascular risk factors and to give guidance and personal advice how to treat risk factors with medication and/or lifestyle.
  Other Names: Disease management; self management; nurse practitioner; internet; risk factors; primary care; vascular diseases
  Arms: internet based intervention

SUMMARY:
The objective of the study is to evaluate the efficacy and cost-effectiveness of an internet based vascular risk factor program on top of usual care compared to usual care alone for treatment of vascular risk factors in patients at high risk for new vascular events.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the efficacy and cost-effectiveness of an internet based vascular risk factor program on top of usual care compared to usual care alone for treatment of vascular risk factors in patients at high risk for new vascular events.

Study design: randomized non-blinded trial Study population: patients in the Rijnstate Hospital Arnhem and the UMC Utrecht, The Netherlands with a recent diagnosis of cerebral, cardiac or peripheral artery disease that entered the risk factor screening programs in these hospitals revealing 2 or more treatable risk factors.

Intervention: After the screening program patients will be randomized to usual care alone or to the internet program on top of usual care. Usual care for risk factor management will be delivered by the medical specialist and/or the general practitioner. Patients randomized to the internet based intervention program are first seen by the nurse practitioner on a regular clinic visit. The internet dossier is than created and explained to the patient. Subsequent contacts between nurse practitioner and patient about risk factor management is mainly by the internet. The nurse practitioner works according to the national guidelines for cardiovascular risk management ('CardioVascular Risico Management 2006') and is supervised by an internist. The study period is 1 year. All patients in both groups ware asked to return to the clinic for a follow up measurement of risk factors after 1 year.

Outcome measures: Primary outcome is the difference in Framingham heart risk score between baseline and after 1 year. As secondary outcome the percentage of patients achieving treatment goals for each risk factor and the average change in the absolute value of each risk factors after 1 year will be used.

Sample size calculation/data analysis: 380 patients. Changes in risk factors (absolute change and fraction of patients achieving treatment goal of each risk factor) at the start and after 1 year and between the groups are tested with independent sample t-test and Chi-square test.

Economic evaluation: The balance between costs and effects of the internet based vascular risk factor management program will be compared to usual care. Using a previously developed cardiovascular disease model incremental cost-utility analyses will be conducted with remaining life expectancy as the relevant time horizon.

ELIGIBILITY:
Inclusion Criteria:

* Participation in a cardiovascular risk screening program
* 2 or more modifiable risk factors not on target:
* SBP > 140 mmHg
* LDL-c > 2.5 mmol/l
* Triglycerides > 1.7 mmol/l
* BMI > 25 kg/m2
* Diabetes Mellitus or fasting glucose > 6.1 mmol/l
* Smoking

Exclusion Criteria:

* No internet access at home
* Unable to read and write Dutch
* Dependent in in daily activities (Ranking score >=3)
* Life expectancy < 2 years or an active malignant disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Framingham heart risk score | 1 year

SECONDARY OUTCOMES:
Percentage of patients achieving treatment goals for each risk factor | 1 year
Additional costs per additional patient achieving treatment goal | 1 year
Cost per life year gained, cost per QALY | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Frank Visseren, MD PhD, Principal Investigator — UMC Utrecht; Yolanda van der Graaf, MD PhD, Study Chair — Julius Center for Health Sciences and Primary Care; Ardine de Wit, MD PhD, Study Chair — Julius Center for Health Sciences and Primary Care; Karin Kaasjager, MD PhD, Study Chair — Rijnstate Hospital Arnhem
Locations (2):
- Netherlands (2):
  - Department of Vascular Medicine UMC Utrecht, Utrecht, Utrecht
  - Rijnstate Hospital, Arnhem

REFERENCES:
- [Background] Goessens BM, Visseren FL, de Nooijer J, van den Borne HW, Algra A, Wierdsma J, van der Graaf Y; SMART Study Group. A pilot-study to identify the feasibility of an Internet-based coaching programme for changing the vascular risk profile of high-risk patients. Patient Educ Couns. 2008 Oct;73(1):67-72. doi: 10.1016/j.pec.2008.06.004. Epub 2008 Jul 18. PMID 18639410
- [Background] Goessens BM, Visseren FL, Sol BG, de Man-van Ginkel JM, van der Graaf Y; SMART Study Group. A randomized, controlled trial for risk factor reduction in patients with symptomatic vascular disease: the multidisciplinary Vascular Prevention by Nurses Study (VENUS). Eur J Cardiovasc Prev Rehabil. 2006 Dec;13(6):996-1003. doi: 10.1097/01.hjr.0000216549.92184.40. PMID 17143135
- [Background] Sol BG, van der Graaf Y, van der Bijl JJ, Goessens BM, Visseren FL. The role of self-efficacy in vascular risk factor management: a randomized controlled trial. Patient Educ Couns. 2008 May;71(2):191-7. doi: 10.1016/j.pec.2007.12.005. Epub 2008 Feb 1. PMID 18242934
- [Background] Sol BG, van der Graaf Y, van der Bijl JJ, Goessens NB, Visseren FL. Self-efficacy in patients with clinical manifestations of vascular diseases. Patient Educ Couns. 2006 Jun;61(3):443-8. doi: 10.1016/j.pec.2005.05.011. Epub 2005 Jul 11. PMID 16009526
- [Background] Sol BG, van der Bijl JJ, Banga JD, Visseren FL. Vascular risk management through nurse-led self-management programs. J Vasc Nurs. 2005 Mar;23(1):20-4. doi: 10.1016/j.jvn.2004.12.003. PMID 15741961
- [Derived] Greving JP, Kaasjager HA, Vernooij JW, Hovens MM, Wierdsma J, Grandjean HM, van der Graaf Y, de Wit GA, Visseren FL. Cost-effectiveness of a nurse-led internet-based vascular risk factor management programme: economic evaluation alongside a randomised controlled clinical trial. BMJ Open. 2015 May 20;5(5):e007128. doi: 10.1136/bmjopen-2014-007128. PMID 25995238
- [Derived] Vernooij JW, Kaasjager HA, van der Graaf Y, Wierdsma J, Grandjean HM, Hovens MM, de Wit GA, Visseren FL; SMARTStudy Group. Internet based vascular risk factor management for patients with clinically manifest vascular disease: randomised controlled trial. BMJ. 2012 Jun 12;344:e3750. doi: 10.1136/bmj.e3750. PMID 22692651